CLINICAL TRIAL: NCT02577471
Title: The Function of Gastrointestinal Tract During Pregnancy and After Delivery
Brief Title: The Function of Gastrointestinal Tract During Pregnancy
Acronym: umpiraskaus
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Other Study IDs: KUH01062012
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Constipation
Keywords: Constipation; pregnancy; delivery
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- During pregnancy: Pregnant ladies filled bowel function questionnaires
- After delivery: ladies within three weeks of delivery filled bowel function questionnaires
- Controls: Non pregnant ladies filled bowel function questionnaires

SUMMARY:
In this prospective study the function of gastrointestinal tract was assessed using constipation questionnaire (Rome criteria and bowel function index).

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained
* pregnancy, delivery
* female non pregnant

Exclusion Criteria:

* no informed consent
* male

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 400 pregnant ladies, 400 ladies who had delivered within three weeks and 200 control ladies who were not pregnant
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Bowel function | one week
  participants filled bowel function questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland